CLINICAL TRIAL: NCT04097665
Title: The Use of Indocyanine Green Angiography to Predict Expanded Flap Viability
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, zantao, Researcher of Plastic and Reconstructive Surgery, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: ICGA
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Necorsis
Keywords: ICGA; necrosis; blood supply; expanded flap
MeSH Terms: conditions — Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with expanded flaps: Patients will undergo tissue expansion. When the expanded flaps are harvested and transplanted, ICGA will be conducted intraoperatively. Meanwhile, the possible area of necrosis will be marked according to clinical experience. And then this area will be further divided into perfusion units (1*1 square centimeter for each). The center of each perfusion unit will be marked as observation point, of which the fluorescence value will be recorded. After 1 week's follow-up postoperatively, the flap tissue will be determined by superimposing digital photography over ICGA imaging results, and the outcome of each observation point will be recorded. By analyzing the fluorescence value and outcome of each observation point, a cut-off point can be further identified to achieve both higher positive and negative predictive value, improving the utility and accuracy of ICGA in predicting the postoperative skin viability of expanded flaps.
  Interventions: Device: indocyanine green angiography

INTERVENTIONS:
Device: indocyanine green angiography — All patients treated with expanded flaps will be assessed by surgeons, and the possible area of necrosis will be marked based on clinical experience. This area will be further divided into perfusion units (1*1 square centimeter for each), and the center of each perfusion unit will be marked. Then all patients will receive ICGA after the complete transfer of flap to the recipient site. For ICGA, a 2ml bolus of indocyanine green (2.5mg/ml) was injected through the patient's intravenous line. The detector/camera of the SPY imaging system should place over the flap at approximately 30cm for fluorescence image acquisition. The fluorescence value will be recorded afterwards.
  Other Names: ICGA

SUMMARY:
It is a prospective and observational trial that designed to evaluate the effect of intraoperative indocyanine green angiography (ICGA) on prediction of postoperative necrosis and other complications in patients treated with expanded flaps.

DETAILED DESCRIPTION:
The lack of suitable soft tissues is a common challenge facing the reconstructive surgeon. Tissue expansion, first described in 1957 by Neumann, is an ingenious technique that can cause body to grow additional skin tissue of similar texture and color to the defect to be repaired and reduce donor site morbidity at the same time. Generally, a silicone balloon expander is inserted under the skin and then gradually filled with saline or carbon dioxide over time, inducing tissue regeneration. Tissue expansion represents one of the major advances in reconstructive surgery and has been widely involved in all kinds of plastic and reconstructive endeavor. In the process of expansion, mechanical stretch also triggers tissue neovascularization and changes in hemodynamic characteristics. These alterations in expanded flap make it challenging to assess flap perfusion and predict postoperative blood flow disorders.

Traditionally, surgeons rely on the clinical experience for determining tissue perfusion, including flap color, capillary refill and pinprick bleeding. However, clinical judgment is highly subjective, difficult to acquire and may be misleading in nonconventional flaps like expanded flaps. Various technologies have been evaluated for perfusion monitoring, including fluorescein angiography, tissue oxygen saturation measurement and thermography. Nevertheless, these are rarely used as routine due to practical limitations, insufficient sensitivity and/or specificity. Recently, Indocyanine Green Angiography (ICGA) has been used for intraoperative evaluation of tissue perfusion. ICGA can give a real-time assessment of flap vascularity and perfusion by intravenously injecting a contrast agent indocyanine green that emits fluorescence when excited by a laser of specific wavelength. Several studies have validated its role in intraoperative evaluation of conventional free and pedicled flap perfusion to aid in surgical decision making and predict postoperative tissue viability. There is obvious difference in hemodynamic characteristics between conventional and expanded flaps so that the conclusion generated from conventional flap study can't be simply extended to expanded flap. In other words, the benefits of ICGA on predicting viability of expanded flaps remains to be validated.

The purpose of this study is to evaluate the effect of intraoperative ICGA on the prediction of flap necrosis in patients underwent tissue expansion. ICGA will be conducted intraoperatively, meanwhile, the possible area of necrosis will be marked according to clinical experience and the fluorescence value of each observation point will be recorded. After 1 week's follow up, the flap viability at each observation point will be assessed by clinical examination. Then, the corresponding fluorescence value will be determined by superimposing digital photography over ICGA imaging results. By analyzing the observation point representing different fate of flap tissue with Logistic regression analysis, ROC curve and area under curve (AUC) can be synthesized by SPSS. A cut-off point can be further identified to achieve both higher positive and negative predictive value, improving the utility and accuracy of ICGA in predicting the postoperative skin viability of expanded flaps.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6-50 years old;
2. Sex: male and female;
3. Undergo expanded flap treatment;
4. Possible to suffer from flap necrosis;
5. Sign the informed consent and are willing to keep following up

Exclusion Criteria:

1. Present or history of significant medical diseases including infectious, renal, cardiovascular, hepatic, hematological and psychiatric diseases;
2. Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for expansion; or history of delayed healing, radiational therapy;
3. Long history of smoking and/or drinking (>5 years) without quit.
4. Iodine allergy; Indocyanine green allergy;
5. Evidence of psychological disorders, no self-awareness and unable to cooperate;
6. Evidence of malignant diseases or unwillingness to participate.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who come to the department of plastic and reconstructive surgery in Shanghai ninth people's hospital and undergo tissue expander treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of necrotic and survival observation points and corresponding intraoperative fluorescence values | 7 days post-operation
  The clinical outcome of each observation point will be assigned as necrosis or survive 7 days post operation. Necrosis includes epidermolysis, partial/superficial necrosis, and full-thickness necrosis. Partial/superficial necrosis is defined as loss of epidermis and partial loss of dermis with no subcutaneous tissue exposure/no requirement for debridement. Full-thickness necrosis is defined as loss of both epidermis and dermis. The number of necrotic and survival observation points will be recorded respectively, and the intraoperative fluorescence value of each point will be backtracked on SPY-Q afterwards.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zan, MD,PhD, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh M, Nuutila K, Kruse C, Robson MC, Caterson E, Eriksson E. Challenging the Conventional Therapy: Emerging Skin Graft Techniques for Wound Healing. Plast Reconstr Surg. 2015 Oct;136(4):524e-530e. doi: 10.1097/PRS.0000000000001634. PMID 26397272
- [Background] Parrett BM, Pomahac B, Orgill DP, Pribaz JJ. The role of free-tissue transfer for head and neck burn reconstruction. Plast Reconstr Surg. 2007 Dec;120(7):1871-1878. doi: 10.1097/01.prs.0000287272.28417.14. PMID 18090749
- [Background] Cherry GW, Austad E, Pasyk K, McClatchey K, Rohrich RJ. Increased survival and vascularity of random-pattern skin flaps elevated in controlled, expanded skin. Plast Reconstr Surg. 1983 Nov;72(5):680-7. doi: 10.1097/00006534-198311000-00018. PMID 6194539
- [Background] Liang X, Huang X, Zhou Y, Jin R, Li Q. Mechanical Stretching Promotes Skin Tissue Regeneration via Enhancing Mesenchymal Stem Cell Homing and Transdifferentiation. Stem Cells Transl Med. 2016 Jul;5(7):960-9. doi: 10.5966/sctm.2015-0274. Epub 2016 Apr 29. PMID 27130223
- [Background] Ghali S, Butler PEM, Tepper OM, Gurtner GC. Vascular delay revisited. Plast Reconstr Surg. 2007 May;119(6):1735-1744. doi: 10.1097/01.prs.0000246384.14593.6e. PMID 17440348
- [Background] Chiu DT, Hu G, Wu J, Rhee S, Rogers L, Gorlick N. Extended rat-ear flap model: a new rodent model for studying the effects of vessel supercharging on flap viability. J Reconstr Microsurg. 2002 Aug;18(6):503-8. doi: 10.1055/s-2002-33322. PMID 12177821
- [Background] Yao ST. Vascular implantation into skin flap: experimental study and clinical application: a preliminary report. Plast Reconstr Surg. 1981 Sep;68(3):404-10. No abstract available. PMID 7267814
- [Background] Moyer HR, Losken A. Predicting mastectomy skin flap necrosis with indocyanine green angiography: the gray area defined. Plast Reconstr Surg. 2012 May;129(5):1043-1048. doi: 10.1097/PRS.0b013e31824a2b02. PMID 22544087
- [Background] Newman MI, Samson MC, Tamburrino JF, Swartz KA. Intraoperative laser-assisted indocyanine green angiography for the evaluation of mastectomy flaps in immediate breast reconstruction. J Reconstr Microsurg. 2010 Sep;26(7):487-92. doi: 10.1055/s-0030-1261701. Epub 2010 Jun 10. PMID 20539977
- [Background] Phillips BT, Lanier ST, Conkling N, Wang ED, Dagum AB, Ganz JC, Khan SU, Bui DT. Intraoperative perfusion techniques can accurately predict mastectomy skin flap necrosis in breast reconstruction: results of a prospective trial. Plast Reconstr Surg. 2012 May;129(5):778e-788e. doi: 10.1097/PRS.0b013e31824a2ae8. PMID 22544108
- [Background] Seifalian AM, Stansby G, Jackson A, Howell K, Hamilton G. Comparison of laser Doppler perfusion imaging, laser Doppler flowmetry, and thermographic imaging for assessment of blood flow in human skin. Eur J Vasc Surg. 1994 Jan;8(1):65-9. doi: 10.1016/s0950-821x(05)80123-9. PMID 8307219
- [Background] Losken A, Styblo TM, Schaefer TG, Carlson GW. The use of fluorescein dye as a predictor of mastectomy skin flap viability following autologous tissue reconstruction. Ann Plast Surg. 2008 Jul;61(1):24-9. doi: 10.1097/SAP.0b013e318156621d. PMID 18580145
- [Background] Li Q, Zan T, Gu B, Liu K, Shen G, Xie Y, Weng R. Face resurfacing using a cervicothoracic skin flap prefabricated by lateral thigh fascial flap and tissue expander. Microsurgery. 2009;29(7):515-23. doi: 10.1002/micr.20640. PMID 19308953
- [Background] Sun BK, Siprashvili Z, Khavari PA. Advances in skin grafting and treatment of cutaneous wounds. Science. 2014 Nov 21;346(6212):941-5. doi: 10.1126/science.1253836. PMID 25414301